CLINICAL TRIAL: NCT05868863
Title: Percutaneous Cementoplasty With or Without Screw Fixation for Bony Pelvis Lesions in Elderly Patients : Feasibility, Safety and Clinical Outcomes.
Brief Title: Percutaneous Cementoplasty With or Without Screw Fixation
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN352023/CHUSTE
Record Dates: First submitted 2023-04-18; First posted 2023-05-22 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Interventional Radiology
Keywords: Cementoplasty; bone pelvic; elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- osteoporotic fractures or neoplastic lesions of the bony pelvis: Patient aged 80 and over suffering from osteoporotic fractures or neoplastic lesions of the bony pelvis treated by percutaneous cementoplasty with or without screw fixation at university hospital center of Saint-Etienne between January 1st 2012 and February 28th 2023 will be included.
  Analysis datas of medical record.
  Interventions: Other: datas of medical record.

INTERVENTIONS:
Other: datas of medical record. — Analysis datas of medical record:
  * Feasibility of the technique
  * Safety of the technique with evaluation by Cardiovascular and Interventional Radiological Society of Europe (CIRSE) scale
  * Analgesic intake before and after the procedure
  * Functional criteria: early rising, walking

SUMMARY:
Bone pathologies such as fragility fractures and neoplastic bone lesions are frequently encountered in rheumatology. When these lesions affect the pelvis, they are responsible both for pain that is sometimes very disabling, but also for significant functional disorders due to their location.

Different methods may be used to treat these lesions. The current challenge is to use less and less invasive techniques such as radio-guided cementoplasty to be able to treat all types of people, especially the most fragile. Among the elderly, the prevalence of these bone pathologies continues to increase due to the aging of the population and the improvement of diagnostic means.

DETAILED DESCRIPTION:
The aim of this study is to retrospectively evaluate the outcome of cementoplasty of the pelvis in people aged 80 and over suffering from osteoporotic fractures or neoplastic lesions of the bony pelvis AND to assess the feasibility, safety and efficiency of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lesion of the bony pelvis treated by percutaneous cementoplasty with or without screw fixation at university hospital center of Saint-Etienne between January 1st 2012 and February 28th 2023

Exclusion Criteria:

* Other interventional treatment at the same time and at the same location

Min Age: 80 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients with lesion of the bony pelvis treated by percutaneous cementoplasty with or without screw fixation at university hospital center of Saint-Etienne between January 1st 2012 and February 28th 2023 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the technique | Months: 3
  Collect from medical records the number of procedures that were completed and performed as theoretically intended.

SECONDARY OUTCOMES:
Safety of the technique by number of adverse events | Months: 3
  collected in the medical record
Number of Analgesic intake before and after the procedure | Months: 3
  collected in the medical record
Analysis Functional criteria: walking | Months: 3
  Collect from medical record the number of patients who can walk before and after the procedure.
Analysis Functional criteria: early rising | Months: 3
  Collect from medical record the number of patients who can rise before and after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain GRANGE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No